CLINICAL TRIAL: NCT06891118
Title: Ultrasound-Guided Stellate Ganglion Block for Refractory Chronic Migraine: a Prospective Evaluation
Brief Title: Stellate Ganglion Blockade for Refractory Chronic Migraine
Acronym: SGB-CM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, Medical doctor, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TABED-2-24-33
Record Dates: First submitted 2025-03-06; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-03

CONDITIONS: Headache, Migraine; Chronic Migraine Headache
Keywords: Migraine, Stellate Ganglion, Nerve Blockade; ultrasonography guided
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, cross-sectional observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SGB blockade patients (Experimental): 18- 65 years of age, diagnosed with chronic migraine in accordance with ICHD-3 criteria, used migraine preventive medication drugs and other interventional algologic treatments that have been applied at least three months ago with insufficient benefit are volunteer patients.
  Interventions: Procedure: Stellate gangion blockade %1 5 mL

INTERVENTIONS:
Procedure: Stellate gangion blockade %1 5 mL — SGB is performed under sterile conditions in the operating room, with the patient's intravenous line established, monitored during the procedure, and ultrasound guidance used simultaneously. The patient is positioned supine, with the neck slightly hyperextended and the head slightly turned to the opposite side. After the skin is cleaned with an antiseptic solution and the probe is sterilized, a linear ultrasound probe is placed transversely at the level of the sixth cervical vertebra (C6).
  The relevant anatomical landmarks, including the internal carotid artery, internal jugular vein, thyroid tissue, longus colli muscle, prevertebral fascia, C6 transverse process (Chassaignac's tubercle), C6 nerve root, and vertebral artery, are visualized. Avoiding vascular structures and thyroid tissue, a 25-gauge 38 mm sterile needle is advanced with a lateral approach using the in-plane technique, ensuring the needle tip is just below the surface of the longus colli m

SUMMARY:
Stellate Ganglion Block (SGB) is a widely used anesthetic technique for treating pain in the head, face, neck, and upper extremities. The procedure involves injecting a local anesthetic into or around the stellate ganglion to temporarily block sympathetic nerve output. It is typically guided by anatomical landmarks, fluoroscopy, or ultrasound, with ultrasound guidance reducing the risk of complications (Yoo 2019).

In migraine patients, repeated ultrasound-guided SGB has been shown to be effective and safe in reducing pain intensity and frequency, as well as improving quality of life by reducing migraine-related disability (Yu-Pain Practice 2023, Hou 2022). It has also demonstrated safety and effectiveness in patients over the age of 65 (Yu-Headache 2023). In clinical practice, ultrasound-guided diagnostic SGB is applied to patients with refractory migraines or chronic headaches who do not respond to pharmacological treatments or peripheral nerve blocks, with positive results leading to weekly repetitions for one month.

Despite studies on the effects of ultrasound-guided SGB in migraine and chronic migraine, there is still no research specifically evaluating its role in treating treatment-resistant chronic migraines after insufficient results from conservative pharmacological treatments and other peripheral nerve blocks. This study aims to evaluate the clinical efficacy of ultrasound-guided SGB in patients with refractory chronic migraines and contribute to the literature. Secondary objectives include assessing its impact on migraine-related disability and monitoring potential side effects and complications.

DETAILED DESCRIPTION:
Migraine is a common neurological disorder, and approximately 8% of migraine patients suffer from chronic migraine (CM), which lasts 15 days or more per month, with at least 8 days of migraine headache characteristics. Chronic migraine (CM) is associated with increased disease burden and socioeconomic disability due to frequent headaches and the lack of pain-free intervals. Therefore, there is a strong need for the effective treatment of migraine and associated symptoms (such as fatigue, sleep disturbances, other pain disorders, other neurological disorders, psychiatric conditions) to reduce disability related to chronic migraine and improve the quality of life. In CM treatment, interventional treatments such as greater occipital nerve (GON) blocks, other peripheral nerve blocks, sphenopalatine ganglion blocks, GON-pulsed radiofrequency (GONPRF), and botulinum toxin injections are commonly applied in pain management practices and in our clinic, when conservative pharmacological treatments fail. Although positive treatment responses have been reported in general, sufficient responses are not always achieved with these interventional treatments in a limited number of patients.

The stellate ganglion is formed by the fusion of the lower cervical and first thoracic sympathetic ganglia and is located in the prevertebral fascia of the C7-T1 vertebrae. Stellate ganglion block (SGB), which involves the injection of a local anesthetic into and around the stellate ganglion to temporarily block sympathetic output, can be beneficial in the treatment of head, face, neck, and upper extremity pain. This procedure is typically performed at the C6 level under anatomical landmarks, fluoroscopy, or ultrasound guidance. Ultrasound is a valuable tool for visualizing soft tissue structures and nerves, guiding the needle insertion, and confirming the spread of the injected material around the target, without exposing doctors and patients to radiation. Concurrent ultrasound-guided SGB helps minimize the risk of serious complications and is considered safer.

SGB is performed under sterile conditions in the operating room, with the patient's intravenous access established, continuous monitoring during the procedure, and real-time ultrasound guidance. Patients are positioned supine, with the neck slightly hyperextended and the head turned slightly to the opposite side. The skin is cleaned with an antiseptic solution, and the probe is covered sterilely. A linear ultrasound probe is placed transversely at the level of the sixth cervical vertebra. Relevant anatomical structures such as the internal carotid artery, internal jugular vein, thyroid tissue, longus colli muscle, prevertebral fascia, C6 transverse process (Chassaignac's tubercle), C6 nerve root, and vertebral artery are visualized. Avoiding vascular structures and thyroid tissue, a 25-gauge, 38-mm sterile needle is advanced laterally using the in-plane technique, with the tip just beneath the prevertebral fascia over the longus colli muscle surface. After confirming the correct position with negative aspiration and 0.5 mL of saline, SGB is performed using 5 mL of 1% lidocaine hydrochloride. For patients with bilateral headaches, SGB is performed on both sides alternately, with a 60-minute interval between applications. For patients with unilateral headaches, SGB is applied to the same side.

Lidocaine hydrochloride is used in a very low dose (50 mg) during unilateral stellate ganglion block. Side effects associated with lidocaine include commonly observed symptoms such as nausea, vomiting, hypotension, hypertension, bradycardia, paresthesia, dizziness, and less commonly, confusion, dysphagia, tremors, tongue numbness, hyperacusis, tinnitus, and rarely allergic or anaphylactic reactions, shock, drowsiness, disorientation, psychosis, irritability, agitation, seizures, convulsions, coma, circumoral paresthesia, blurred and double vision, transient amaurosis, cardiac disturbances like heart block, cardiovascular collapse, arrhythmias, and myocardial depression, as well as respiratory and chest issues such as dyspnea, bronchospasm, apnea, respiratory depression, and respiratory arrest. Long-term use can lead to temporary liver dysfunction, and high concentrations may affect the central nervous system and cardiovascular system, leading to loss of consciousness, convulsions, excessive muscle activity, hypotension, bradycardia, arrhythmias, or even cardiac arrest.

Recent studies have shown that SGB can be beneficial in the treatment of migraine and chronic migraine. An observational study reported that ultrasound-guided SGB was effective in reducing the intensity and frequency of pain in migraine patients and could reduce migraine-related disability, thereby improving the patients' quality of life. A retrospective observational study of 52 migraine patients aged 65 and older, who underwent ultrasound-guided SGB, showed that SGB treatment could reduce headache intensity, frequency, duration, and the need for additional treatments, and that it could be a safe and effective intervention in elderly patients with migraine. Another retrospective observational study reported that ultrasound-guided SGB was an effective and safe treatment for chronic migraine patients, with repeated SGB sessions providing benefit.

In our clinic, we apply diagnostic SGB under ultrasound guidance in patients who do not respond to GONB, other peripheral nerve blocks, GONPRF, sphenopalatine ganglion blocks, and in those whose chronic migraine-related headaches and disability negatively impact daily living activities. We repeat the procedure weekly for patients who report a positive response, over a period of one month.

Although there are limited studies evaluating the effects of ultrasound-guided SGB in the treatment of migraine and chronic migraine, there is still no study specifically assessing the role of SGB in treating resistant chronic migraine in cases where conservative pharmacological treatment, as well as GON and/or other peripheral nerve blocks, GONPRF, and sphenopalatine ganglion blocks, have not yielded sufficient results. The primary aim of our study is to evaluate the clinical efficacy of ultrasound-guided stellate ganglion block in patients with resistant chronic migraine and contribute to the literature. The secondary aims are to assess the impact of ultrasound-guided SGB on migraine-related disability and to observe any potential side effects and complications associated with the treatment.

ELIGIBILITY:
Inclusion Criteria:

18- 65 years of age, diagnosed with chronic migraine in accordance with ICHD-3 criteria, used migraine preventive medication drugs and other interventional algologic treatments that have been applied at least three months ago with insufficient benefit are volunteer patients.

Exclusion Criteria:

* Migraine according to ICHD-3 criteria has a history of primary headache other than migraine, migraine preventive interventional treatment within the last 3 months and/or botulinum toxin A, nonpharmacological treatment (acupuncture, ozone, cognitive behavioral therapy, etc.), injection infection at the site, pregnancy or suspected pregnancy, known allergy to local anesthetic drugs with a history of malignancy or cranial/cervical surgery, bleeding-coagulation disorder or oral anticoagulants, comorbid diseases that may cause headache (uncontrolled hypertension, intracranial lesions), with diseases that may prevent compliance with treatment (psychiatric disorder, dementia) and patients who did not accept the planned interventional treatment were excluded from the study.

will be released.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 months
  With VAS, a 10-point VAS score of 0 is no pain and 10 is the highest intensity pain that can be endured

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Privacy.

REFERENCES:
- See also: Yu B, Zhang W, Zhao C, Xing Y, Meng L, Luo F. Effectiveness, safety, and predictors of response to ultrasound-guided stellate ganglion blockades for the treatment of patients with chronic migraine: A retrospective and observational study. Pain Pract.2023 — https://pubmed.ncbi.nlm.nih.gov/31337167/
- See also: Yu B, Hou S, Xing Y, Jia Z, Luo F. Ultrasound-guided stellate ganglion block for the treatment of migraine in elderly patients: A retrospective and observational study. Headache. 2023; 63:763-770. doi:10.1111/head.14537. — https://pubmed.ncbi.nlm.nih.gov/31337167/